CLINICAL TRIAL: NCT00132405
Title: Randomized, Double-Blind, Placebo-Controlled Study to Determine the Effectiveness and Safety of ALGRX 3268 0.5 Mg/20 Bar at the Back of the Hand in Pediatric Subjects
Brief Title: Study of ALGRX 3268 for Needlestick Pain in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlgoRx Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3268-2-002-1
Record Dates: First submitted 2005-08-15; First posted 2005-08-22 (Estimated); Last update posted 2005-10-10 (Estimated); Status verified 2005-08

CONDITIONS: Pain
Keywords: Needlestick pain; Venipuncture pain; Procedural pain
MeSH Terms: conditions — Pain; Pain, Procedural

INTERVENTIONS:
Drug: ALGRX 3268

SUMMARY:
Minor needlestick procedures often cause significant pain and distress in children, yet interventions to reduce pain are used infrequently. ALGRX 3268 is a novel, single-use, prefilled, needle-free dispenser that immediately delivers powdered lidocaine into the epidermis and provides local analgesia in 2 to 3 minutes. The purpose of this prospective, randomized, double-blind, and placebo-controlled trial is to determine the efficacy and tolerability of ALGRX 3268 in children aged 3 to 18 years undergoing venipuncture. The trial will enroll a total of 306 children aged 3 to 18 years scheduled to undergo venipuncture of the back of the hand at a single study center.

DETAILED DESCRIPTION:
ALGRX 3268 (previously known as PowderJect® Dermal Lidocaine) is a system for needle-free, pain-free epidermal injection of lidocaine powder that provides local anesthesia within 3 minutes to provide painless needle or catheter insertion for blood drawing. ALGRX 3268 is a single use disposable system, incorporating a drug cassette and gas cylinder into a single hand held device, with a button to actuate the system. This is a single center, randomized, double-blind, placebo (sham) controlled, single dose, parallel group study in pediatric subjects scheduled to undergo venipuncture. Three age groups are enrolled: 3-7 years, 8-12 years, and 13-18 years. Within each age group, subjects are randomized to receive ALGRX 3268 0.5 mg/20 bar or pressure matched placebo. Two to 3 minutes after administration of study treatment at the back of the hand, venipuncture is performed with either a needle/Vacutainer®, needle/syringe or "butterfly," at the discretion of the investigator. Subjects aged 3-7 are asked to rate the pain of venipuncture using the Wong-Baker FACES Pain Rating Scale, anchored at 0 for "no hurt" and 5 for "hurts worst." Subjects in oldest age group complete a 100 mm visual analogue scale (VAS), anchored at 0 for "no pain" and at 100 for "extreme pain." Subjects in the middle group used both the Wong-Baker FACES scale and the VAS to rate the pain of venipuncture. Safety ratings of skin are completed 15, 30, and 60 minutes after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient children of either gender who were to undergo venipuncture at the back of the hand
* Children must have had sufficient cognitive skills to identify faces depicting extremes of pain on the Wong-Baker FACES Pain Rating Scale (ages 3-12) and/or the extremes of pain on a 100 mm VAS (ages 8-18).
* Ages 3 to 7 years; 8 to 12 years; and 13 to 18 years, inclusive
* Consent forms must have been approved by the appropriate Institutional Review Board (IRB). Signed informed consent must have been granted by the parent or legal guardian and assent to participate should have been sought (either verbally or in writing) from each child.
* In females of childbearing potential, who in the judgment of the investigator or designee were sexually active, a negative urine pregnancy test must have been documented prior to enrollment. A negative urine pregnancy test was required in all teenage girls over the age of 14 years. Surgically sterile females did not require a pregnancy test.

Exclusion Criteria:

* Previous history of allergic reactions to any local anesthetic
* Any medical condition or instability that, in the judgment of the investigator, might have adversely impacted the conduct of the study and the collection of data
* Subjects in whom the investigator determined that venipuncture could not be accomplished cleanly
* Active local infection or other skin pathology on the dorsum of the hand
* Subjects with tattoos, surgical scars, ports, implantable devices or a skin condition that may have interfered with placement of study treatment or skin site assessments
* Female subjects who were pregnant or lactating; females who planned to become pregnant; females with a positive serum or urine pregnancy test; females of childbearing potential who were not using adequate contraception.
* Prior participation in an ALGRX 3268 study
* Venipuncture at the proposed site within the prior two weeks (longer if bruising was apparent)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260
Dates: Start 2004-05; Study Completion 2004-09

PRIMARY OUTCOMES:
Subject's assessment of the pain of venipuncture following administration of study treatment

SECONDARY OUTCOMES:
Parents are asked to assess their child's level of pain of venipuncture on a 100 mm visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: William Zempsky, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States